CLINICAL TRIAL: NCT05492123
Title: Randomized Phase II Study to Evaluate Induction Nivolumab-Ipilimumab, Followed by Nivolumab With Chemoradiotherapy Versus Chemoradiotherapy for Advanced Cervical Cancer
Brief Title: Nivolumab-ipilimumab and Chemoradiation for Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Bristol-Myers Squibb (Industry); Brava (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRAVA- Cervical - SGPP 5031-21
Record Dates: First submitted 2022-07-22; First posted 2022-08-08 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-01

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Uterine Cervical Neoplasms; Nivolumab; Ipilimumab; Chemoradiation; Anti-PD1; Anti-PDL1; Anti-CTLA4; Immunotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Nivolumab; Injections; Ipilimumab; Chemoradiotherapy

STUDY DESIGN:
Intervention Model Description: Prospective randomized trial, stratified by center, disease stage and type of radiation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Chemoradiation (Active Comparator): Traditional radiation therapy with a target of 45 Gy in 25 1.8Gy fractions with concurrent weekly cisplatin 40mg/m2/week or carboplatin AUC 2/week
  Interventions: Radiation: Chemoradiation
- Immunotherapy (Experimental): 4 cycles of induction therapy with nivolumab 1mg/kg and ipilimumab 3mg/kg every 3 weeks followed by traditional radiation therapy with a target of 45 Gy in 25 1.8Gy fractions with concurrent weekly cisplatin 40mg/m2/week (or carboplatin AUC 2/week) with concurrent nivolumab 240mg every 2 weeks.
  Interventions: Drug: Nivolumab 40 mg in 4 ml Injection; Drug: Ipilimumab 200 MG in 40 ML Injection; Radiation: Chemoradiation

INTERVENTIONS:
Drug: Nivolumab 40 mg in 4 ml Injection — Nivolumab 1mg/kg every 3 weeks for 4 cycles prior to radiation and 240mg every 2 weeks with concurrent radiation
  Other Names: Opdivo
  Arms: Immunotherapy
Drug: Ipilimumab 200 MG in 40 ML Injection — Ipilimumab 3mg/kg every 3 weeks for 4 cycles prior to radiation
  Other Names: Yervoy
  Arms: Immunotherapy
Radiation: Chemoradiation — Radiation to a dose of 45Gy over 25 1.8Gyfractions and brachytherapy with concurrent weekly cisplatin 40mg/m2/w or carboplatin AUC 2/w
  Other Names: Cisplatin-based chemoradiation

SUMMARY:
A total of 112 patients with locally advanced cervical cancer will be randomized 1:1 to standard therapy with cisplatin-based chemoradiation or nivolumab-ipilimumab induction followed by cisplatin-based chemoradiation. The primary outcome will be 3-year disease-free survival.

DETAILED DESCRIPTION:
Patients with adenocarcinoma or squamous cell carcinoma of the cervix, FIGO Stage IB2-IB3 node positive or Stage IIB-IVA will be randomized to conventional cisplatin-based chemo-radiation or to 4 cycles of induction immunotherapy with nivolumab 1mg/kg and ipilimumab 3mg/kg every 3 weeks, followed by cisplatin chemo-radiation with concurrent nivolumab 240mg every 2 weeks. Primary outcome will be 3-year progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Female participants older than 18 years
* Documented evidence of cervical adenocarcinoma or squamous carcinoma FIGO Stage IB2-IB3 node positive or Stage IIB-IVA
* No prior chemotherapy, immune checkpoint inhibitors or radiotherapy for cervical cancer
* WHO/ECOG performance status of 0-1
* At least 1 lesion, not previously irradiated, that qualifies as a RECIST 1.1 Target Lesion at baseline.

Exclusion Criteria:

* Diagnosis of small cell (neuroendocrine) histology cervical cancer
* Intent to administer a fertility-sparing treatment regimen
* Undergone a previous hysterectomy
* Evidence of metastatic disease per RECIST 1.1 including lymph nodes ≥15 mm (short axis) above the L1 cephalad body or outside the planned radiation field.
* History of allogeneic organ transplantation
* Active or prior documented autoimmune or inflammatory disorders
* Uncontrolled intercurrent illness
* History of another primary malignancy and active primary immunodeficiency
* Patients with active infection

Laboratory values that fall into:

1. WBC count (WBC) < 2000/μL ;
2. Neutrophil count < 1500/μL;
3. Platelet count < 100 x 103/μL;
4. Hemoglobin level < 9.0 g/dL;
5. Serum creatinine > 1.5 x upper limit of normal (ULN) unless creatinine clearance is

   ≥ 40 mL/min (measured or calculated using the Cockcroft-Gault formula);
6. Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT): > 3.0 x ULN;
7. Total bilirubin > 1.5 x ULN (except participants with Gilbert Syndrome who must have a total bilirubin level of < 3.0 x ULN);
8. Any positive test result for hepatitis B virus or hepatitis C virus that indicates the presence of the virus, for example, positive Hepatitis B surface antigen (HBsAg, Australia antigen) or Hepatitis C antibodies (anti- HCV) positive (unless the HCV-RNA is negative).

   * Participants with a condition requiring systemic treatment or with corticosteroids (>10 mg daily of a prednisone equivalent) or other immunosuppressive drugs within 14 days of initiating study treatment.
   * Pregnant or breastfeeding woman

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
3-year progression-free survival | 3 years
  No evidence of disease recurrence/regrowth after 3 years of follow-up

SECONDARY OUTCOMES:
3-year overall survival | 3 years
  Rate of survival 3 years after the end of chemoradiation
Objective response rate | 90 days after the end of chemoradiation
  RECIST response
Response duration | Through study completion, an average of 3 year
  Time from maximum response to disease progression
To evaluate health related quality of life (HRQoL): defined as the change from baseline of disease-related symptoms and quality of life of patients undergoing treatment Nivolumab-ipilimumab and Chemoradiation for Cervical Cancer | Baseline (time from screening - before starting treatment) and at the end of treatment (56 days after the last dose of radiotherapy).
  Evaluate health related quality of life using the instrument EORTC QLQ-C30 v3 based on European Organization for Research and Treatment of Cancer (EORTC). The EORTC QLQ-C30 v3 questionnaire, consisting of 30 questions covering 15 domains, divided into three distinct scales: state scale global health and quality of life (it has only one domain, global health measure); functional scale (physical function, role performance, emotional function, cognitive function and social function domains); and symptom scale (fatigue, nausea and vomiting, pain, dyspnea, insomnia, loss of appetite, constipation, diarrhea and financial difficulties). The scores on each scale range from 0 - 100. The global and functional health scales indicate better quality of life as their score approaches 100. For the symptoms scale, the analysis is inverse, with better performance for quality of life when the scores approach the score minimum (zero).
Evaluate health related quality of life using supplemental cervical cancer module (EORTC CX24) to evaluate patients submitted to treatment with Nivolumab-ipilimumab and Chemoradiation for Cervical Cancer. | Baseline (time from screening - before starting treatment) and at the end of treatment (56 days after the last dose of radiotherapy).
  The EORTC - CX24 questionnaire contains 24 questions, divided into three multiple-item scales and six single-item scales, of which 11 refer to symptoms (questions 31-37, 39 and 41-43), three about body image. (questions 45-47), four questions on sexual/vaginal function (questions 50-53), one on lymphedema (question 38), one for evaluation of peripheral neuropathy (question 40), one for evaluation of menopausal symptoms (question 44) ), one on sexual concerns (question 48), one on sexual activity (question 49) and one on sexual pleasure (question 54). The answers are transformed into a score from 0 - 100 and calculated separately for each scale.
Treatment-related toxicity | Through study completion, an average of 3 year
  Treatment-related toxicity according to CTCAE version 4.0 (Common Toxicity Criteria for Adverse Events )

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Maluf, MD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (14):
- Brazil (14):
  - CRIO -Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Clinica AMO, Salvador, Estado de Bahia
  - Hospital das Clinicas da UFMG, Belo Horizonte, Minas Gerais
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Multi Oncoclinicas Recife, Recife, Pernambuco
  - Hospital São Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Universidade Federal de Roraima, Boa Vista, Roraima
  - CEPON - Florianópolis, Florianópolis, Santa Catarina
  - Hospital de Amor, Barretos, São Paulo
  - Hospital De Base de São José do Rio Preto - CIP São José, São José do Rio Preto, São Paulo
  - INCA - Instituto Nacional do Cancer, Rio de Janeiro
  - AC Camargo Cancer Center, São Paulo
  - Hospital Municipal Vila Santa Catarina, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chemoradiotherapy for Cervical Cancer Meta-Analysis Collaboration. Reducing uncertainties about the effects of chemoradiotherapy for cervical cancer: a systematic review and meta-analysis of individual patient data from 18 randomized trials. J Clin Oncol. 2008 Dec 10;26(35):5802-12. doi: 10.1200/JCO.2008.16.4368. Epub 2008 Nov 10. PMID 19001332
- [Background] Naumann RW, Hollebecque A, Meyer T, Devlin MJ, Oaknin A, Kerger J, Lopez-Picazo JM, Machiels JP, Delord JP, Evans TRJ, Boni V, Calvo E, Topalian SL, Chen T, Soumaoro I, Li B, Gu J, Zwirtes R, Moore KN. Safety and Efficacy of Nivolumab Monotherapy in Recurrent or Metastatic Cervical, Vaginal, or Vulvar Carcinoma: Results From the Phase I/II CheckMate 358 Trial. J Clin Oncol. 2019 Nov 1;37(31):2825-2834. doi: 10.1200/JCO.19.00739. Epub 2019 Sep 5. PMID 31487218
- [Background] Santin AD, Deng W, Frumovitz M, Buza N, Bellone S, Huh W, Khleif S, Lankes HA, Ratner ES, O'Cearbhaill RE, Jazaeri AA, Birrer M. Phase II evaluation of nivolumab in the treatment of persistent or recurrent cervical cancer (NCT02257528/NRG-GY002). Gynecol Oncol. 2020 Apr;157(1):161-166. doi: 10.1016/j.ygyno.2019.12.034. Epub 2020 Jan 7. PMID 31924334